CLINICAL TRIAL: NCT01119235
Title: A Phase 1, Open Label Study To Investigate The Pharmacokinetics Of Multiple Doses Of PF-04531083 Tablets In Healthy Volunteers
Brief Title: A Study To Observe The Performance Of A Tablet Form Of PF-04531083 As Evidenced By The Concentration Of PF-04531083 In The Blood With Time Following Oral Administration To Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1351005
Record Dates: First submitted 2010-04-19; First posted 2010-05-07 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Pain
Keywords: Pharmacokinetics; tablet performance; healthy volunteers; open label
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: PF-04531083 (Active Comparator)
  Interventions: Drug: PF-04531083
- Cohort 2: PF-04531083 (Active Comparator)
  Interventions: Drug: PF-04531083

INTERVENTIONS:
Drug: PF-04531083 — Dosed as a tablet in 100mg strengths. Dosage in the first cohort will be 300mg twice daily for 3 days followed by 200mg twice daily for 11 days
  Arms: Cohort 1: PF-04531083
Drug: PF-04531083 — Dosed as a tablet in 100mg strengths. Dosage in this optional second cohort will be optimised based on the data arising from Cohort 1
  Arms: Cohort 2: PF-04531083

SUMMARY:
A new tablet form of PF-04531083 has been manufactured. Previously the compound was administered as a solution/suspension to healthy volunteers. This study will investigate the pharmacokinetics of PF-044531083 in tablet form and compare with the pharmacokinetics obtained, with the same dosing regimen, with the solution/suspension.

ELIGIBILITY:
Inclusion Criteria:

* Young
* Healthy volunteers

Exclusion Criteria:

* Elderly volunteers
* Patients with any existing medical conditions considered likely to impinge on study execution

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
concentration of PF-04531083 in blood just before dosing on the 8th day of the study | Days 1 and 8 of the study

SECONDARY OUTCOMES:
pharmacokinetic parameters derived from the plasma concentration versus time profile of PF-04531083 following single and multiple dosing. AUCtau, Cmax, Tmax will be calculated. | Days 1, 8 and 14 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1351005&StudyName=A%20Study%20To%20Observe%20The%20Performance%20Of%20A%20Tablet%20Form%20Of%20PF-04531083%20As%20Evidenced%20By%20The%20Concentration%20Of%20PF-04531083%20In%20The%20Blood%20W